CLINICAL TRIAL: NCT06465342
Title: PROSPECTIVE MULTICENTER OBSERVATIONAL CLINICAL INVESTIGATION OF LUTEIN USE BY SCLERAL IONTOPHORESIS IN PATIENTS WITH STAGE 3 AGE-RELATED MACULAR DEGENERATION (AMD)
Brief Title: LUTEIN BY SCLERAL IONTOPHORESIS IN PATIENTS WITH STAGE 3 AGE-RELATED MACULAR DEGENERATION (AMD)
Status: Not yet recruiting | Type: Observational
Sponsor: OFFHEALTH S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: IONTO/06/2023
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: DML Stage 3

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the clinical investigation is to evaluate the performance, safety and degree of tolerability resulting from the use of the iontophoresis medical device in adult subjects diagnosed with AMD stage 3 (AREDS classification) in one or both eyes.

DETAILED DESCRIPTION:
Lutein is a dietary carotenoid which, together with its isomer zeaxanthin, is the main component of the macular pigment of the retina.

Clinical studies have shown that prolonged oral lutein supplementation is safe and is associated with a reduction in the risk of progression from early to advanced stages of Age-Related Macular Degeneration (AMD). However, patient compliance, due to daily oral intake of lutein tablets for a prolonged period of life, is still limited. Additionally, an obstacle to oral supplementation is the variable absorption of lutein through the digestive route.

An iontophoresis method for conveying substances into the eye has been known for some time and already used in the treatment of keratoconus. In this case the substance conveyed is Riboflavin.

A medical device is now available with the following intended use: to combat all oxidative pathologies of the retina and macula, and in particular in the prevention of AMD and in the management of the patient during the evolution of the pathology.

The device consists of an iontophoresis system with scleral applicator and an ophthalmic liquid lutein solution, both of which have already obtained the CE mark. The system therefore includes a generator called K-IONO (CE in class IIa) and a kit called IONTORETINA, which includes a sterile 2 ml vial of lutein (CE in class IIb), the forward and return electrode . which consists of a scleral iontophoresis applicator and an ophthalmic liquid solution of lutein. The topical application of lutein has the advantage of improving the patient's compliance with lutein supplementary therapy compared to oral intake of the carotenoid; Furthermore, in situ application would allow high (therapeutic) concentrations of lutein to be reached in the macular area in a very short period of time (hours) compared to oral intake (months). Publicly available clinical data on scleral iontophoresis or lutein supplementation have not demonstrated any safety-related adverse events and at the same time have demonstrated a reduction in the cumulative risk of progression of AMD from intermediate to advanced stages of the disease.

The objective of the clinical investigation is to evaluate the performance, safety and degree of tolerability resulting from the use of the iontophoresis medical device in adult subjects diagnosed with AMD stage 3 (AREDS classification) in one or both eyes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (male or female) aged ≥ 55 years;
* Subject able to provide Informed Consent, in compliance with good clinical practice and current legislation (i.e. subject able to understand the full nature and purpose of the clinical investigation, including any risks and side effects);
* Subject with age-related macular degeneration (AMD) category 3 in one or both eyes classified according to the criteria reported by "Age-Related Eye Disease Study (AREDS)" based on clinical manifestations:
* Subject in good general health;
* Manifest spherical equivalent refraction between +4.0 diopters (D) and - 4.0 D;
* Best corrected visual acuity (BCVA) for glasses ≤ 0.1 LogMAR;
* Intraocular pressure (IOP) ≤ 20 mmHg;
* Subject willing to perform a consistent dietary plan, dietary supplement, and medication regimen throughout the study;
* Subject able to comply with the requirements of the clinical investigation plan, according to the Investigator;
* Subjects available for the entire period of the study;
* Subjects able to cooperate with the Investigator;
* Subjects able to meet the requirements of the entire clinical investigation;
* Subject who qualifies for treatment with Iontoretina according to the approved indication;
* Subject who, in the opinion of the Investigator, will draw benefit from this treatment.

Exclusion Criteria:

* Ocular surgery or other type of invasive intervention within the previous 3 months (of any type, including laser surgery and intravitreal injections) performed on the study eye;
* Lesions, scars, or abrasions of the ocular components present in the eye under study;
* Dense opacities of the ocular components of the study eye;
* Implantation of intraocular lenses (IOLs) in the study eye;
* Congenital malformations in the study eye;
* Medical history of ocular hypertension and glaucoma, macular pucker, optic neuropathy, diabetic retinopathy, dry eye syndrome, etc. (limited to the study eye);
* Ocular infection or acute or chronic inflammation of the study eye (for example: Herpes simplex infections, corneal virus infections, bacterial, viral or fungal conjunctivitis, tuberculosis and mycosis of the eye, purulent and herpetic blepharitis, stye, uveitis, dacryocystitis);
* Concomitant treatments (topical and/or systemic) with medications, dietary supplements, and/or medical devices known to have effects on the eye; (digitoxin, quinoline, chlorpromazine, tamoxifen, thiazide diuretics);
* Lutein or zeaxanthin supplementation or any supplementation or with the intention of impacting eye health within the last 4 weeks prior to the screening visit;
* Known or potential allergy or hypersensitivity and/or history of allergic reactions to any of the components of the medical device or other chemically closely related substances;
* Subject suffering from type I diabetes, or with a previous case of stroke;
* Subject suffering from uncontrolled hypertension and heart disease that, in the opinion of the Investigator, does not allow participation in the study or could compromise the results;
* Evidence of severe or uncontrolled systemic disease or any other significant disorder, which in the opinion of the Investigator does not allow participation in the study or could impair the results;
* Subject smoker (more than 20 cigarettes per day);
* Significant alcohol consumption: more than 2 drinks per day;
* Women of childbearing potential will be excluded from participation in the study if they meet any of the following conditions:
* pregnant;
* intend to become pregnant during the study treatment period;
* breastfeeding, or unwilling to use birth control methods that can be considered highly effective for the entire duration of the study;
* Concomitant hormone replacement therapy for menopause.
* Participation in another clinical study within the previous 90 days;
* Subject unable to follow clinical investigation procedures and follow-up visits;
* Any other medical condition that, in the opinion of the Investigator, could affect participation in the clinical investigation or impair its results.

Ages: 55 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects (male and female), suffering from stage 3 AMD over 55 years of age. 80 eyes belonging to subjects of both sexes who will be recruited with competitive enrollment between the sites involved in the clinical investigation.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-06-12 (Estimated); Primary Completion 2025-09-12 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
BCVA changes | 12 months
  Changes in best distance-corrected visual acuity (BCVA) at the End of Study Visit compared to baseline.

SECONDARY OUTCOMES:
BCVA changes | 3, 4, 5 and 6 monhs
  Changes in best distance-corrected visual acuity (BCVA) at scheduled controls (Visit 3, Visit 4, Visit 5, and Visit 6) compared to baseline